CLINICAL TRIAL: NCT06677866
Title: Effectiveness of Cooperative Group Therapy in Adolescents With Fragile X Syndrome (FXS) and in Adolescents With Autism Spectrum Disorder (ASD)
Brief Title: Group CBT in Adolescents With Fragile X Syndrome and in Adolescents With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Paolo Alfieri, medical doctor, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2850_OPBG_2022
Record Dates: First submitted 2024-10-23; First posted 2024-11-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Fragile X Syndrome (FXS); Autism Spectrum Disorder
Keywords: intellectual disability; adaptive functioning; quality of life; rare genetic syndrome; Cognitive Behavioral Therapy; CBT; fragile x syndrome; autism spectrum disorder; neuropsychology
MeSH Terms: conditions — Fragile X Syndrome; Autism Spectrum Disorder; Intellectual Disability | interventions — Cognitive Behavioral Therapy; Waiting Lists

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study is conducted by four main professionals: the neuropsychiatrist principal investigator (Dr. Paolo Alfieri) responsible for the FXS treatment group; the neuropsychiatrist (Dr. Giovanni Valeri) responsible for the ASD treatment group; the cognitive behavioral therapist performing the intervention with the FXS treatment group (Dr. Alice Federica Maria Montanaro) and the cognitive behavioral therapist performing the intervention with the ASD treatment group (Dr. Laura Casula).
  The two neuropsychiatrists conducting the clinical evaluation of the severity of the disorder and the presence of changes following the intervention (using the CGI-S scale) remain blind to treatment allocation during the trial and analyses until the conclusion of the study. Furthermore, the evaluating psychologists (who are different from the two therapists performing the intervention) and a speech therapist perform blinded assessments at T0-T1-T2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASD-CGT- Treatment group (ASD-CGT) (Experimental): Group of adolescents with ASD that perform the intervention at the beginning of the study (ASD-CGT)
  Interventions: Behavioral: Cognitive behavioral therapy
- FXS- Waiting List group (FXS-WL) (Other): Group of adolescents with FXS that perform the intervention once that the sections with the first group are ended (FXS-WL)
  Interventions: Other: Waiting List
- FXS- CGT- Treatment group (FXS-CGT) (Experimental): Group of adolescents with FXS that perform the intervention at the beginning of the study (FXS-CGT)
  Interventions: Behavioral: Cognitive behavioral therapy
- ASD- Waiting List group (ASD-WL) (Other): Group of adolescents with ASD that perform the intervention once that the sections with the first group are ended (ASD-WL)
  Interventions: Other: Waiting List

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Cooperative Group Therapy (CGT) is a cognitive-behavioral group therapy based on the theoretical and practical principles of the Cooperative Parent-Mediated Therapy model [Valeri et al., 2020].
  The goal of CGT is to promote the following core skills: Pragmatics, Executive Functions, and Cooperative Interactions. The CGT program consists of 15 sessions over a total duration of 6 months: 12 group therapy sessions with adolescents and 3 sessions with their parents. Each session focuses on a specific topic and lasts between 90 and 120 minutes.
  The CGT therapist is a psychotherapist with a cognitive-behavioral orientation who utilizes evidence.-based strategies to enhance pragmatic, socio-conversational skills, cognitive flexibility, emotional regulation, and cooperative interactions. The CGT intervention is conducted by two cognitive-behavioral psychotherapists specialized respectively in the treatment of FXS and ASD.
  Arms: ASD-CGT- Treatment group (ASD-CGT); FXS- CGT- Treatment group (FXS-CGT)
Other: Waiting List — The Waiting List (WL) is a control group in which participants who do not receive the experimental treatment are placed on a waiting list to receive the intervention after the active treatment group has completed it. In the case of the WL, the CGT intervention is carried out after at least 6 months to allow the patients in the first group to complete the treatment cycle. This approach enables a comparison between a group of treated patients and a group of patients who have not yet been treated, while still allowing the latter to access the treatment at a later stage.
  Arms: ASD- Waiting List group (ASD-WL); FXS- Waiting List group (FXS-WL)

SUMMARY:
Fragile X Syndrome (FXS) is a rare genetic syndrome, caused by a mutation in the FMR1 gene located on the X chromosome. It is considered the leading hereditary cause of intellectual disability (ID) and the primary cause of Autism Spectrum Disorder (ASD) due to a single gene-mutation. Many individuals with FXS exhibit symptoms overlapping with those of ASD, including difficulties in social-communication skills, challenges in peer relationships, restricted and repetitive behaviors/interests and deficits in adaptive functioning. Both in ASD and FXS, individuals with greater deficits in executive functions, socio-pragmatic, and socio-relational skills also demonstrate lower adaptive functioning and, consequently, reduced autonomy/independence throughout the life course and greater severity of the disorder.

Among empirically validated treatments recommended by National and International Guidelines for the treatment of ASD, cognitive-behavioral and psychosocial interventions have been shown to improve some aspects of ASD, such as core symptoms, emotional-behavioral disturbances, adaptive skills, and quality of life. Currently, it appears that cognitive-behavioral therapies, which include psychoeducation programs, are particularly appropriate for ASD, with greater efficacy for group interventions compared to individual ones. Regarding FXS, despite the well-established knowledge of the cognitive-behavioral phenotype and the clear need for scientifically validated programs, research on intervention strategies remains quite limited.

Considering the similarities between ASD and FXS and the need for standardized interventions, the present research project aims to conduct an RCT to evaluate the feasibility of Cooperative Group Therapy (CGT) in two different groups of adolescents with ASD and FXS. The decision to target the intervention to adolescents is due to the few clinical studies on this age group, which is a crucial target since, in FXS, there is often a plateau or reversal of intellectual and adaptive development after the age of 10, and in adolescents with ASD, the development and complexity of social, pragmatic skills, and executive functions are crucial for good adaptive functioning and a basic quality of life. Te main hypothesis is that CGT could contribute to the reduction of severity illness and in the enhancement of socio-communicative skills.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder affecting approximately 1% of the global population, characterized by early onset, difficulties in communication and reciprocal social interaction, and associated with unusually restricted and repetitive behaviors and interests.

Fragile X Syndrome (FXS) is a rare genetic syndrome affecting about 1 in 4.,000 males and 1 in 8.,000 females, caused by a mutation in the FMR1 gene located on the X chromosome. It is considered the leading hereditary cause of intellectual disability (ID) and the primary cause of ASD due to a mutation in a single gene.

Research shows that many individuals with FXS exhibit symptoms overlapping with those of ASD, including difficulties in social-communication skills, challenges in peer relationships, restricted and repetitive behaviors/interests, and deficits in adaptive functioning. In both syndromes, individuals with greater deficits in executive functions, socio-pragmatic, and socio-relational skills also demonstrate lower adaptive functioning and, consequently, reduced autonomy/independence throughout the life course and greater severity of the disorder.

Among empirically validated treatments recommended by National and International Guidelines for the Treatment of Autism, cognitive-behavioral and psychosocial interventions have been shown to improve some aspects of ASD, such as core symptoms, emotional-behavioral disturbances, adaptive skills, and quality of life. Currently, it appears that cognitive-behavioral therapies, which include psychoeducation programs, are particularly appropriate for ASD, with greater efficacy for group interventions compared to individual ones. However, a very recent meta-analysis of Conrad and colleagues (2021) highlighted that there are currently only 30 RCTs (Randomized Clinical Trials) on ASD and that most of these studies have been conducted in a limited geographical area, with few studies in Europe. Regarding FXS, despite the well-established knowledge of the cognitive-behavioral phenotype and the clear need for scientifically validated programs, research on intervention strategies remains quite limited. In a 2011 systematic review, Moskowitz and Carr analyzed 31 studies investigating the effectiveness of behavioral treatment in FXS and pointed out that most of them were conducted with limited methodological rigor. Indeed, their review revealed that the examined interventions employed various behavioral strategies, often using a single patient per technique, making it difficult to draw conclusions about individual techniques. The lack of empirically validated cognitive-behavioral intervention models remains a significant issue for all clinicians working with individuals with FXS and ASD. Consequently, parents continue to rely on intervention methods whose clinical effectiveness has not been tested, monitored, or replicated through studies with valid methodological rigor. As a result, there is an undeniable need to develop new interventions: a) conducted with methodological rigor (RCTs), b) applicable across different age groups, and c) structured, empirically measurable, and replicable.

In 2020, Valeri and colleagues conducted the first European RCT to assess the clinical effectiveness of Cooperative Parent-Mediated Therapy (CPMT) in preschool children with Autism, showing that CPMT is effective in improving socio-communication skills, core ASD symptoms, and in reducing parental stress related to dysfunctional parent-child interactions.

Subsequently, in 2021, Alfieri and colleagues conducted a study to verify the efficacy of CPMT in treating socio-communicative deficits in children with FXS and Williams Syndrome, demonstrating that the use of a parent-mediated intervention, theoretically founded and utilizing ECEN strategies (Evolutive and Naturalistic Behavioral Interventions), results in significant improvement in socio-communicative-relational skills even in these populations.

Additionally, Montanaro and coll. in 2020 performed a study to examine the efficacy of Corp-osa-Mente (CoM), a combined neuropsychological and cognitive behavioral group therapy (nCBT) tailored on young adults and targeting the different clinical manifestations of FXS through a unified approach. Results indicated an improvement in participants' psychopathological symptoms, cognitive abilities, and general adaptive behavior. However the study faced different methodological issues, such as the absence of standardized measures. Therefore, additional methodologically rigorous studies were required to substantiate these initially promising findings.

Based on these encouraging results in children and adults with FXS, the present research project aims to conduct an RCT to evaluate the clinical efficacy and feasibility of Cooperative Group Therapy (CGT) in two different groups of adolescents with ASD and FXS. The decision to target the intervention to adolescents is due to the few clinical studies on this age group, which is a crucial target since, in FXS, there is often a plateau or reversal of intellectual and adaptive development after the age of 10, and in adolescents with ASD, the development and complexity of social, pragmatic skills, and executive functions are crucial for good adaptive functioning and a decent quality of life. Specifically, the primary goal is the reduction of the mean score on the Global Clinical Impression - Severity Scale (CGI-S), which measures the severity of the disorder, after treatment compared to baseline. Pre- and post-treatment evaluations of cognitive and adaptive profiles will also be conducted, and standardized questionnaires will be administered, with results used as secondary endpoints (e.g., Social Responsiveness Scale, SRS; Behavior Rating Inventory of Executive Functioning, BRIEF; Vineland Adaptive Behavior Scales -II, VABS-II; Multidimensional Anxiety Scale for Children-II, MASC II; Child Behavior Checklist, CBCL; Conners' Parent Rating Scale, CPRS; Quality of Life Scale, QoLS; Parenting Stress Index, PSI).

ELIGIBILITY:
FXS group:

Inclusion Criteria

* Clinical diagnosis of FXS confirmed by genetic testing.
* Age between 13 and 19 years.
* Language skills compatible with group intervention (verbal language at sentence level).
* Impairment in adaptive functioning measured by VABS II < 70.
* Informed consent for participation and data processing provided by parents. Exclusion Criteria
* Severe visual or hearing impairments.
* Diagnosis of epilepsy or a history of seizures requiring medication.
* Participation in other non-pharmacological treatments.
* Changes in pharmacological therapy within the last 3 months.
* Presence of medical problems or behaviors that could interfere with group activities, as measured by the Autism Behavior Checklist (ABC) (ABC Irritability Scale < 18).
* IQ < 40 measured by the Leiter third edition (Leiter 3)
* Severe adaptive functioning, measured by VABS II < 20.

ASD group:

Inclusion Criteria

* Clinical diagnosis of Autism Spectrum Disorder (ASD) confirmed by ADOS-2 and ADI-R interviews.
* Age between 13 and 19 years.
* Language skills compatible with group intervention (verbal language at sentence level).
* Impairment in adaptive functioning measured by VABS II < 70.
* Informed consent for participation and data processing provided by parents.

Exclusion Criteria

* Severe visual or hearing impairments.
* Identification of specific genetic abnormalities or presence of known genetic syndromes associated with ASD (e.g., TSC, FXS, 22q11, 16p11.2, Rett Syndrome).
* Diagnosis of epilepsy or a history of seizures requiring medication.
* Participation in other non-pharmacological treatments.
* Changes in pharmacological therapy within the last 3 months.
* Presence of medical problems or behaviors that could interfere with group activities, as measured by the Autism Behavior Checklist (ABC) (ABC Irritability Scale < 18).
* IQ < 40 measured by the Leiter third edition (Leiter 3)
* Severe adaptive functioning, measured by VABS II < 20.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Global Clinical Impression - Severity Scale (CGI-S) | 6 months
  - Clinical improvement: Clinical Global Impression - Severity scale Clinical Global Impression - Severity scale is a 7-point scale used to measure baseline severity of patients (Higher scores indicate more severe patient)

SECONDARY OUTCOMES:
Clinical Global Impression - Improvement scale (CGI-I) | 6 months
  Changes in Clinical Global Impression - Improvement scale (CGI-I) is a 7-point scale used to measure improvement after treatment. Higher scores indicate more severe symptoms.
Child Behavior Checklist 6-18 (CBCL 6-18) | 6 months
  Changes in Behavioral and emotional problems as measured by the Child Behavior Checklist (CBCL) 6-18. Higher scores indicate severe problems. According to the ASEBA Assessment Data Manager (ADM), t-scores of Syndrome Scales, DSM-Oriented Scale and 2007 Scales from 67 to 70 fall in the borderline range, while t-scores above 70 in the clinical range; concerning the Total Problem, Internalizing, and Externalizing Scale, t-scores of 60 to 63 delineate the borderline range, while t-scores above 63 delineate the clinical range. Changes in Adaptive Level
Total Scale and the Subdomains of the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) | 6 months
  Changes in the adaptive functioning of adolescents measured by the Total Scale and the Subdomains of the Vineland Adaptive Behavior Scales, Second Edition (VABS-II). Scores are expressed in standard scores (mean 100, Standard deviation 15). Higher scores indicate better functioning.
Parenting Stress Index Short Form (PSI- SF) | 6 months
  Changes in the parenting stress as measured by the Parenting Stress Index Short Form, Total Score and Subscales scores. Scores are expressed in percentile (from 5th to 100th). Higher scores indicate higher level of stress.
Pediatric Quality of Life- Family Impacts | 6 months
  Changes in the Pediatric Quality of Life- Family Impact. Higher scores indicate higher quality of life.
Multidimensional Anxiety Scale for Children-II (MASC-II) | 6 months
  Changes in the levels of anxiety as measured by the Multidimensional Anxiety Scale for Children-II (MASC-II). Higher scores indicate severe problems. 60-64 slightly elevated, 65-69 elevated, ≥70 very elevated.Changes in the behavioral and attentional symptomatology across multiple settings
Conners' Parent Rating Scale (CPRS) | 6 months
  Changes in behavioral and attentional symptomatology measured by the Conners' Parent Rating Scale (CPRS). Higher scores indicate severe problems. >64 borderline >70 clinical.
Social Responsiveness Scale (SRS) | 6 months
  Changes in social responsiveness measured by the Social Responsiveness Scale (SRS) Total Scores and Subtests scores. Higher scores indicate severe problems. >64 borderline >70 clinical.
Behavior Rating Inventory of Executive Functioning second edition (BRIEF II) | 6 months
  Changes in the executive functioning measured by the Total Score and the subtests scores of Behavior Rating Inventory of Executive Functioning second edition (BRIEF II), parent report form. Higher scores indicate severe problems. >64 borderline >70 clinical.
Kiddie Schedule for Affective Disorders and Schizophrenia Present and Lifetime Version (KSADS-PL) | 6 months
  Change from baseline in the KSADS diagnosis. The K-SADS-PL for DSM-5 is a semi-structured diagnostic interview that ascertains both lifetime and current diagnostic episodes in children and adolescents
Children's Global Assessment Scale | 6 months
  Changes in the Children's Global Assessment Scale (CGAS). CGAS is a clinician rating of overall adaptive functioning during the previous month for children and adolescents between 4 to 16 years of age. CGAS scores are rated on a 100-point scale, with 1 being the most impaired and 100 being least impaired, and descriptors for each 10-point interval such that each 10-point interval defines a range of children's functioning in all areas of their life. CGAS scores were secondary outcome measures. The Change in Children's Global Assessment Scale (CGAS) measures level of general functioning on a 100 point scale - 1 (needs constant supervision) to 100 (superior functioning). Every 10 points global functioning moves to the next category.
Children's Communication Checklist - Second Edition (CCC-2) | 6 months
  Changes in the communication profiles as measured by the Children's Communication Checklist - Second Edition (CCC-2). Ths is a test that assesses the presence of communicative problems of a pragmatic nature that are difficult to assess with traditional tests. It includes the following subscales: Eloquence, Syntax, Semantics, Coherence, Inappropriate beginning, Stereotyped language, Use of context, Non-verbal communication, Social relations, Interests. Using these subscales, two global scores can be calculated, the Global Communication Score (GCC) and the Social Interaction Deviance Index (SIDI). A scaled score of 6 or higher is considered a normal score for the subscales. A GCC score of 55 or less is considered clinically significant and indicating a possible communication disorder. Conversely, negative overall SIDI means that there is significant discrepancy between language and social interaction abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Alfieri, MD, PhD, Principal Investigator — Bambino Gesù Children's Hospital; Stefano Vicari, MD, clinical professor, Study Chair — Bambino Gesù Hospital and Research Institute
Locations (1):
- Bambino Gesù Children's Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Valeri G, Casula L, Menghini D, Amendola FA, Napoli E, Pasqualetti P, Vicari S. Cooperative parent-mediated therapy for Italian preschool children with autism spectrum disorder: a randomized controlled trial. Eur Child Adolesc Psychiatry. 2020 Jul;29(7):935-946. doi: 10.1007/s00787-019-01395-5. Epub 2019 Sep 23. PMID 31549310
- [Result] Alfieri P, Scibelli F, Casula L, Piga S, Napoli E, Valeri G, Vicari S. Cooperative Parent-Mediated Therapy in Children with Fragile X Syndrome and Williams Beuren Syndrome: A Pilot RCT Study of a Transdiagnostic Intervention-Preliminary Data. Brain Sci. 2021 Dec 23;12(1):8. doi: 10.3390/brainsci12010008. PMID 35053752
- [Result] Montanaro FAM, Alfieri P, Caciolo C, Spano G, Bosco A, Vicari S. Effects of a combined neuropsychological and cognitive behavioral group therapy on young adults with Fragile X Syndrome: An explorative study. Res Dev Disabil. 2024 Nov;154:104839. doi: 10.1016/j.ridd.2024.104839. Epub 2024 Sep 26. PMID 39332280